CLINICAL TRIAL: NCT03999047
Title: Validation of the Screening Instrument: PRISMA-7 for Frailty Among +75 Year Old Danes Still in Need of Physical Training When They Are Sent Home After a Hospital Stay
Brief Title: Validation of the Screening Instrument: PRISMA-7 for Frailty Among Elderly Hospitalized Danes
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Region Zealand (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Ellen Holm, Consultant, Region Zealand
Other Study IDs: REG-070-2017; 707462 (Other: Institute of Healtresearch)
Record Dates: First submitted 2019-06-16; First posted 2019-06-26 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Frailty Syndrome
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: PRISMA score — Screening for frailty using PRISMA-7

SUMMARY:
The questionnaire PRISMA-7 was originally developed to assess frailty in community dwelling adults. The questionnaire was translated into the Danish language. This instrument was used to screen for frailty among elderly patients (75+) sent home from Nykøbing Falster Hospital after a hospital admission during the period 31. May 2017 until December 31st, 2018. PRISMA results were used to categorize each individula as frail or non-frail. The register of PRISMA results was merged with national registers on use of health serviced in order to investigate if increasing PRISMA score was associated with increasing use of health services.

DETAILED DESCRIPTION:
Data from PRISMA scores were registered in an EasyTrial database. This database is recognized by the regional health authorities as a safe system to store individual health data. All use of the EasyTRial database is logged. The merging of data from the local EasyTRial database with data from national registries on use of health services and on mortality was permitted by the Danish National Health Data protection authorities.

ELIGIBILITY:
Inclusion Criteria:

* 75 years old persons being returned from hospital after a hospital admission and in need of further physical rehabilitation in the community

Exclusion Criteria:

Not able to give informed consent or if necessary not having a relative that can give informed consent

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Persons 75 years old og older who have been staying in hospital and are in need physical rehabilitation in the municipality when they are sent home from hospital.
Sampling Method: Non-Probability Sample
Enrollment: 1050 (Actual)
Dates: Start 2019-06-16 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | 6 months after PRISMA-7 screening
  Mortality
Morbidity | 6 months after Prisma-7 screening
  Morbidity will be measured by registering Hospital admissions and use of general practitioner

SECONDARY OUTCOMES:
Use of other health services | 6 months before PRISMA-7 screening
  Home help, rehabilitation services in the municipality
Morbidity | 6 months after PRISMA-7 screening
  Morbidity will be measured by registering hospital admissions and use og general practitioner

CONTACTS AND LOCATIONS:
Overall Officials: Ellen A Holm, MD, Principal Investigator — Region Sjælland
Locations (1):
- Nykøbing Falster Hospital, Nykøbing Falster, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Turner G, Clegg A; British Geriatrics Society; Age UK; Royal College of General Practioners. Best practice guidelines for the management of frailty: a British Geriatrics Society, Age UK and Royal College of General Practitioners report. Age Ageing. 2014 Nov;43(6):744-7. doi: 10.1093/ageing/afu138. PMID 25336440
- [Background] Hebert R, Durand PJ, Dubuc N, Tourigny A; PRISMA Group. Frail elderly patients. New model for integrated service delivery. Can Fam Physician. 2003 Aug;49:992-7. PMID 12943358
- [Background] Raiche M, Hebert R, Dubois MF. PRISMA-7: a case-finding tool to identify older adults with moderate to severe disabilities. Arch Gerontol Geriatr. 2008 Jul-Aug;47(1):9-18. doi: 10.1016/j.archger.2007.06.004. Epub 2007 Aug 27. PMID 17723247
- [Background] Braun T, Gruneberg C, Thiel C. German translation, cross-cultural adaptation and diagnostic test accuracy of three frailty screening tools : PRISMA-7, FRAIL scale and Groningen Frailty Indicator. Z Gerontol Geriatr. 2018 Apr;51(3):282-292. doi: 10.1007/s00391-017-1295-2. Epub 2017 Aug 9. PMID 28795247
- [Background] Hoogendijk EO, van der Horst HE, Deeg DJ, Frijters DH, Prins BA, Jansen AP, Nijpels G, van Hout HP. The identification of frail older adults in primary care: comparing the accuracy of five simple instruments. Age Ageing. 2013 Mar;42(2):262-5. doi: 10.1093/ageing/afs163. Epub 2012 Oct 28. PMID 23108163
- [Background] Lynge E, Sandegaard JL, Rebolj M. The Danish National Patient Register. Scand J Public Health. 2011 Jul;39(7 Suppl):30-3. doi: 10.1177/1403494811401482. PMID 21775347
- [Background] Andersen JS, Olivarius Nde F, Krasnik A. The Danish National Health Service Register. Scand J Public Health. 2011 Jul;39(7 Suppl):34-7. doi: 10.1177/1403494810394718. PMID 21775348
- [Background] Kildemoes HW, Sorensen HT, Hallas J. The Danish National Prescription Registry. Scand J Public Health. 2011 Jul;39(7 Suppl):38-41. doi: 10.1177/1403494810394717. PMID 21775349

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-20): https://cdn.clinicaltrials.gov/large-docs/47/NCT03999047/Prot_SAP_000.pdf